CLINICAL TRIAL: NCT05720793
Title: A Clinical Trial to Evaluate the Safety and Tolerability of Fecal Microbiota Transplantation in a Population With Obsessive-compulsive Disorder
Brief Title: A Clinical Trial of Fecal Microbiota Transplantation in a Population With Obsessive-compulsive Disorder
Acronym: FOCUSED
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Valerie Taylor (Other)
Collaborators: Nimble Science Ltd. (Industry); University of Calgary (Other)
Responsible Party: Sponsor-Investigator, Valerie Taylor, MD, Phd, FRCPC, Professor, Department Head, University of Calgary
Organization: University of Calgary (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIM-FMT/OCD-2022
Record Dates: First submitted 2023-01-26; First posted 2023-02-09 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; Microbiome; FMT; Gut bacteria
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT capsule + SIMBA Capsule (Experimental): adults with OCD who are being treated with an approved first line treatment for OCD medication will be assigned to receive FMT capsules as an adjunct treatment.
  Interventions: Combination Product: FMT Capsule + SIMBA Capsule

INTERVENTIONS:
Combination Product: FMT Capsule + SIMBA Capsule — Participants in this arm will receive FMT capsules in addition to their usual treatment. participants will also be administered SIMBA sample collection capsules.

SUMMARY:
Obsessive-compulsive disorder (OCD) is a psychiatric condition marked by recurrent intrusive thoughts (obsessions) and ritualistic behaviors aimed at reducing distress (compulsions). While there exist a number of medications to treat this illness, half of those who need them either do not respond or can not tolerate current medications because of side effects. Therefore, there is an urgent need to develop new ways to treat this illness. One of the areas being explored as a potential option is based on what is now known as a strong link between the bacteria that live in our gut and the brain. Research has shown that a fecal transplant of the gut bacteria from healthy donors is able to improve health outcomes for people with depression and the investigators now want to expand this into OCD, given a known link between this condition and bacterial infection. To do this the investigators will use both the standard methods of bacterial identification via stool analysis, which looks at large bowel changes, and compare it to the Small Intestine Microbiome Aspiration (SIMBA) system, a small capsule that when swallowed allows a fluid sample to be collected from the participants' small intestine. This work will help the investigators assess the benefits of fecal transplant in OCD, and more importantly, identify how transplant changes the system, utilizing a novel technology to move the field forward.

ELIGIBILITY:
Inclusion Criteria:

* Adults who have a primary diagnosis of OCD
* on a stable appropriate dose of (SSRI) treatment for at least 12 weeks prior to Baseline
* insufficient response to current SSRI treatment indicated by persistence of symptoms.

Exclusion Criteria:

* Participant meets Diagnostic criteria for substance use, eating disorder, schizophrenia, or schizoaffective disorder
* Suicidality
* regular intake of antibiotics, prebiotics, or probiotics
* Clinically diagnosed with IBD, Crohn's disease, Ulcerative colitis, or Celiac disease
* Immune suppression
* intestinal obstruction
* Oropharyngeal dysphagia or other swallowing disorder
* < 2 bowel movements per week
* Breastfeeding, pregnant or seeking to get pregnant during the course of this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 0-13 weeks
  Reported Adverse events
Toronto Side Effects Scale (TSES) | 0-13 weeks
  Changes in the Toronto Side Effects Scale (TSES). TSES a 32-item instrument used to evaluate the incidence, frequency, and severity of the central nervous system (CNS), gastrointestinal (GI), and sexual side effects.

SECONDARY OUTCOMES:
Global function/overall improvement (Quick Inventory of Depressive Symptomatology-Self-Report (QIDS)) | 0-13 weeks
  Quick Inventory of Depressive Symptomatology-Self-Report (QIDS). is a 16-item questionnaire that rates depression symptoms via self-assessment. Toral score is calculated but summing the scores of each of the 16 different questions. 0-5 Normal, 6-10 mild depression, 11-15 Moderate depression, 16-20 Severe depression and >21 is considered very severe depression.
Global function/overall improvement (The General Anxiety Disorder-7 scale (GAD-7)) | 0-13 weeks
  The General Anxiety Disorder-7 scale (GAD-7). The 7-item tool is used to screen and assess for generalized anxiety. Score 0-4: Minimal Anxiety, Score 5-9: Mild Anxiety, Score 10-14: Moderate Anxiety and Score greater than 15: Severe Anxiety
Global function/overall improvement (Positive and Negative Affect Schedule (PANAS)) | 0-13 weeks
  Positive and Negative Affect Schedule (PANAS). The PANAS is a self-report questionnaire that consists of two 10-item scales and measures both positive and negative emotions for participants. The total score is calculated by finding the sum of the 10 positive items, and then the 10 negative items. Scores range from 10 - 50 for both sets of items. higher score indicates more positive or negative affect respectively.
Global function/overall improvement (Patient Health Questionnaire-9(PHQ9)) | 0-13 weeks
  Patient Health Questionnaire-9(PHQ9). The PHQ9 is used for screening and measuring the severity of depressive symptoms. The total score is the sum the numbers of all the checked responses under each heading. Cut off scores are: 0 - 4 None, 5 - 9 Mild, 10 - 14 Moderate, 15 - 19 Moderately Severe and 20 - 27 Severe.
OCD symptoms (Y-BOCS) | 0-13 weeks
  Yale-Brown Obsessive Compulsive Scale (Y-BOCS). Total scores range from 0 to 40. 0-7 indicates subclinical symptoms, 8-15 mild symptoms, 16-23 moderate symptoms, 24-31 severe symptoms and 32-40 extreme symptoms
OCD symptoms (TOCS) | 0-13 weeks
  Toronto Obsessive-Compulsive Scale (TOCS). TOCS is a 21 item self-reported questionnaire that assesses several major symptom dimensions in OCD. A total score is calculated by adding each score of the 21 items, and dimension scores are calculated by averaging the sum of item scores within each dimension.
Next generation fecal, Urine, Blood and saliva sequencing | 0-13 weeks
  analysis of Fecal, urine, blood and saliva samples

CONTACTS AND LOCATIONS:
Overall Officials: Valere Taylor, MD,PhD,FRCPC, Principal Investigator — Professor, Head of Department
Locations (1):
- University of Calgary, TRW building, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
We will also share our results via the "Gut Microbiota for Health Experts exchange", an online community where experts in this field share news, innovation and information on topics pertaining to the gut microbiota (www.gutmicrobiotaforhealth.com). This organization has over 10 000 online members and a large social media presence. Manuscripts will be published in scientific journals

REFERENCES:
- [Background] Wlodarska M, Kostic AD, Xavier RJ. An integrative view of microbiome-host interactions in inflammatory bowel diseases. Cell Host Microbe. 2015 May 13;17(5):577-91. doi: 10.1016/j.chom.2015.04.008. PMID 25974300
- [Background] O'Hara AM, Shanahan F. The gut flora as a forgotten organ. EMBO Rep. 2006 Jul;7(7):688-93. doi: 10.1038/sj.embor.7400731. PMID 16819463
- [Background] Gorkiewicz G, Moschen A. Gut microbiome: a new player in gastrointestinal disease. Virchows Arch. 2018 Jan;472(1):159-172. doi: 10.1007/s00428-017-2277-x. Epub 2017 Dec 14. PMID 29243124
- [Background] Liu HN, Wu H, Chen YZ, Chen YJ, Shen XZ, Liu TT. Altered molecular signature of intestinal microbiota in irritable bowel syndrome patients compared with healthy controls: A systematic review and meta-analysis. Dig Liver Dis. 2017 Apr;49(4):331-337. doi: 10.1016/j.dld.2017.01.142. Epub 2017 Jan 21. PMID 28179092
- [Background] Zhong L, Shanahan ER, Raj A, Koloski NA, Fletcher L, Morrison M, Walker MM, Talley NJ, Holtmann G. Dyspepsia and the microbiome: time to focus on the small intestine. Gut. 2017 Jun;66(6):1168-1169. doi: 10.1136/gutjnl-2016-312574. Epub 2016 Aug 3. No abstract available. PMID 27489239
- [Background] Grace E, Shaw C, Whelan K, Andreyev HJ. Review article: small intestinal bacterial overgrowth--prevalence, clinical features, current and developing diagnostic tests, and treatment. Aliment Pharmacol Ther. 2013 Oct;38(7):674-88. doi: 10.1111/apt.12456. Epub 2013 Aug 20. PMID 23957651
- [Background] Ghoshal UC, Shukla R, Ghoshal U. Small Intestinal Bacterial Overgrowth and Irritable Bowel Syndrome: A Bridge between Functional Organic Dichotomy. Gut Liver. 2017 Mar 15;11(2):196-208. doi: 10.5009/gnl16126. PMID 28274108
- [Background] Luna RA, Foster JA. Gut brain axis: diet microbiota interactions and implications for modulation of anxiety and depression. Curr Opin Biotechnol. 2015 Apr;32:35-41. doi: 10.1016/j.copbio.2014.10.007. Epub 2014 Nov 21. PMID 25448230
- [Background] Camilleri M. Probiotics and irritable bowel syndrome: rationale, putative mechanisms, and evidence of clinical efficacy. J Clin Gastroenterol. 2006 Mar;40(3):264-9. doi: 10.1097/00004836-200603000-00020. PMID 16633134
- [Background] Desbonnet L, Garrett L, Clarke G, Bienenstock J, Dinan TG. The probiotic Bifidobacteria infantis: An assessment of potential antidepressant properties in the rat. J Psychiatr Res. 2008 Dec;43(2):164-74. doi: 10.1016/j.jpsychires.2008.03.009. Epub 2008 May 5. PMID 18456279
- [Background] Eutamene H, Bueno L. Role of probiotics in correcting abnormalities of colonic flora induced by stress. Gut. 2007 Nov;56(11):1495-7. doi: 10.1136/gut.2007.124040. PMID 17938427
- [Background] Gareau MG, Jury J, MacQueen G, Sherman PM, Perdue MH. Probiotic treatment of rat pups normalises corticosterone release and ameliorates colonic dysfunction induced by maternal separation. Gut. 2007 Nov;56(11):1522-8. doi: 10.1136/gut.2006.117176. Epub 2007 Mar 5. PMID 17339238
- [Background] Sullivan A, Nord CE. Probiotics and gastrointestinal diseases. J Intern Med. 2005 Jan;257(1):78-92. doi: 10.1111/j.1365-2796.2004.01410.x. PMID 15606379
- [Background] Girard SA, Bah TM, Kaloustian S, Lada-Moldovan L, Rondeau I, Tompkins TA, Godbout R, Rousseau G. Lactobacillus helveticus and Bifidobacterium longum taken in combination reduce the apoptosis propensity in the limbic system after myocardial infarction in a rat model. Br J Nutr. 2009 Nov;102(10):1420-5. doi: 10.1017/S0007114509990766. Epub 2009 Jun 29. PMID 19563693
- [Background] Logan AC, Katzman M. Major depressive disorder: probiotics may be an adjuvant therapy. Med Hypotheses. 2005;64(3):533-8. doi: 10.1016/j.mehy.2004.08.019. PMID 15617861
- [Background] Rao AV, Bested AC, Beaulne TM, Katzman MA, Iorio C, Berardi JM, Logan AC. A randomized, double-blind, placebo-controlled pilot study of a probiotic in emotional symptoms of chronic fatigue syndrome. Gut Pathog. 2009 Mar 19;1(1):6. doi: 10.1186/1757-4749-1-6. PMID 19338686
- [Background] Messaoudi M, Lalonde R, Violle N, Javelot H, Desor D, Nejdi A, Bisson JF, Rougeot C, Pichelin M, Cazaubiel M, Cazaubiel JM. Assessment of psychotropic-like properties of a probiotic formulation (Lactobacillus helveticus R0052 and Bifidobacterium longum R0175) in rats and human subjects. Br J Nutr. 2011 Mar;105(5):755-64. doi: 10.1017/S0007114510004319. Epub 2010 Oct 26. PMID 20974015
- [Background] Dickerson FB, Stallings C, Origoni A, Katsafanas E, Savage CL, Schweinfurth LA, Goga J, Khushalani S, Yolken RH. Effect of probiotic supplementation on schizophrenia symptoms and association with gastrointestinal functioning: a randomized, placebo-controlled trial. Prim Care Companion CNS Disord. 2014;16(1):PCC.13m01579. doi: 10.4088/PCC.13m01579. Epub 2014 Feb 13. PMID 24940526